CLINICAL TRIAL: NCT01013623
Title: A Phase III, Randomized Trial of Surgical Resection With or Without BCG Versus Best Medical Therapy as Initial Treatment in Stage IV Melanoma
Brief Title: Stage IV Surgery Versus Best Medical Therapy
Acronym: STG4SURG
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Lack of accrual, lack of continued funding.
Sponsor: Saint John's Cancer Institute (Other)
Collaborators: Melanoma Research Alliance (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MORD-STG4SURG-0409; 3P01CA012582-35S1 (NIH)
Record Dates: First submitted 2009-11-12; First posted 2009-11-16 (Estimated); Last update posted 2012-09-26 (Estimated); Status verified 2012-09

CONDITIONS: Stage IV Resectable Melanoma
Keywords: melanoma; stage IV; resectable; surgery; medical therapy
MeSH Terms: conditions — Melanoma | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Best Medical Therapy (Active Comparator): The best medical therapy group will not initially undergo surgery, but will be treated with the therapy that medical oncologists or surgeons feel is best for the patient. This treatment may include standard or experimental therapies.
  Interventions: Other: best medical therapy
- Surgery Alone (Active Comparator): The surgery alone group will undergo complete resection (surgical removal) of all known disease, if possible. After surgery, patients will be followed regularly and monitored for disease recurrence.
  Interventions: Procedure: Surgery
- Surgery + BCG (Active Comparator): The Surgery + BCG group will first have a complete resection (surgical removal) of all known disease, if possible. After recovery from surgery, two doses of BCG will be given two weeks apart. Each dose is given as 8 separate injections into the skin (called intradermal injections).
  Interventions: Procedure: Surgery plus 2 adjuvant doses of BCG

INTERVENTIONS:
Procedure: Surgery — surgical resection to remove all known disease
  Arms: Surgery Alone
Procedure: Surgery plus 2 adjuvant doses of BCG — Patients in the surgical resection + BCG arm will have an additional two visits to receive BCG. The first dose of BCG will be given no earlier than 4 weeks after surgery, and the second BCG dose will follow 2 weeks later. The actual doses are determined by the patient's pre-study tuberculin-reactivity status. Patients with a pre-study PPD induration of ≥10 mm will be given half the normal dose of BCG. Those with PPD induration of ≥20 mm will be given 25% of the normal dose.
  Arms: Surgery + BCG
Other: best medical therapy — Patients randomized to the Best Medical Therapy arm will decide on a course of medical therapy based on what the patient's medical oncologists feels is best for the patient. Best systemic medical therapy may include clinical trials of new agents or standard non-protocol treatments. Patients who progress on the best medical treatment arm may switch to a different medical therapy or, if still appropriate, may receive surgery.
  Arms: Best Medical Therapy

SUMMARY:
This study will establish the role of surgical versus nonsurgical approaches in patients whose melanoma has spread to distant sites. Results will help clinicians develop a standardized initial approach that prolongs survival and optimizes quality of life. Results also will indicate whether Bacillus Calmette-Guerin (BCG) postoperative immunotherapy significantly improves the outcome of patients treated with surgery.

DETAILED DESCRIPTION:
This study is designed to examine the impact of surgical resection versus medical therapy as initial treatment therapy for patients with Stage IV melanoma. Surgical resection is thought to be efficacious in highly selected patients with solitary metastases, but not in patients with multiple sites of metastases. Even in those with solitary metastases, there is considerable debate among major melanoma centers over whether undergoing initial systemic medical therapy prior to surgical resection should be preferred to initial surgical resection upon Stage IV diagnosis. According to Dr. Dan Coit, Co-leader of the Melanoma Disease Management Team at Memorial Sloan Kettering Cancer Institute in New York, a trial of initial medical therapy is their standard approach on the multidisciplinary melanoma service even for patients with solitary distant metastases (personal communication, 15 Dec 2009).

Many who favor upfront medical therapy believe that delay before surgical resection may avoid unnecessary surgery by identifying patients who progress early due to the outgrowth of occult metastases at multiple sites, which may make the patient unresectable.

This is a Phase III, randomized, international, multicenter study of metastasectomy with or without BCG versus best medical therapy as initial therapy in Stage IV melanoma. This study has three arms: surgical resection plus BCG as an immune adjuvant, surgical resection plus observation, and best medical therapy (BMT). Since no systemic medical therapy has been demonstrated to be superior to DTIC and multiple new therapies are being evaluated, the choice as to what constitutes best medical therapy will be determined by the individual investigator based on the standard of care for systemic medical therapy at that particular multicenter site. Best systemic medical therapy may include clinical trials of new agents or standard non-protocol treatments (e.g., DTIC or Temodar according to the standard of care at the multi-center site).

Patients who progress on the best medical treatment arm may switch to a different medical therapy or, if appropriate, have surgical therapy; similarly, surgery patients may have additional surgical resection or receive medical therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients must provide informed written consent for participation.
* At least 18 years of age
* Have a minimum life expectancy (excluding melanoma) of 5 years.
* All known disease must be surgically resectable in the opinion of a participating surgeon.
* Must have a histologic diagnosis of Stage IV melanoma arising from a primary cutaneous site or visceral metastasis from an unknown primary site and be within 4 months of initial stage IV diagnosis.
* Up to 3 visceral organs involved
* Up to 6 lesions allowed
* Must have ECOG performance status of 0 or 1.
* Must be in good general health with no serious co-morbid illness. Good clinical judgment must be exercised in careful selection of patients who are candidates for surgical resection of distant metastases.
* Laboratory values within 30 days of randomization:

  1. WBC >3,000/mm3
  2. Lymphocytes >800/mm3
  3. Platelets >100,000/mm3
  4. Creatinine <2.0 mg/dL
  5. Bilirubin <2.0 mg/dL
  6. Alkaline phosphatase < 2X upper limit of normal (ULN)
  7. SGOT < 2X ULN
  8. SGPT < 2X ULN
  9. LDH < 1.5X ULN

Exclusion Criteria:

* Unresectable metastatic disease or more than 4 months since stage IV diagnosis.
* Brain or bone metastatic sites.
* History of primary uveal or mucosal melanoma.
* Another concomitant diagnosis that limits life expectancy to less than 5 years.
* Chronic immunosuppression due to inherited, acquired or iatrogenic immune defect. This includes active HIV, hepatitis, or use of immunosuppressive medications as a component of anti-rejection therapy for organ transplant, as treatment for an autoimmune disease.
* More than 3 involved visceral organ sites or more than 6 metastatic lesions.
* Psychiatric disorder or organic brain syndrome that might preclude participation in the protocol.
* Diagnosis of other malignancy in the past 5 years except adequately treated low grade malignancies such as basal cell carcinoma, cutaneous squamous cell carcinoma, carcinoma-in-situ of the cervix, or other neoplasm that will not limit life expectancy to less than 5 years.
* Serious cardiac, gastrointestinal, hepatic or pulmonary disease that would make surgical resection high-risk.
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2009-11; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Overall survival | 3 interim analyses will be conducted when 75, 148, and 217 events (deaths) have occurred. The final analysis will be conducted when all 284 expected events have occurred.
  Defined as time from randomization to death from any cause

SECONDARY OUTCOMES:
Time to progression of initial metastatic sites (progression-free survival) | 3 interim analyses will be conducted when 75, 148, and 217 primary events have occurred. The final analysis will be conducted when all 284 expected events have occurred.
  For this study, PFS is defined as the time from randomization to disease recurrence at initial metastatic site in patients rendered disease-free by surgery, or time from randomization to RECIST-defined progression of target lesions in patients receiving best medical therapy or those having residual disease following surgery.
Melanoma-specific survival | 3 interim analyses will be conducted when 75, 148, and 217 recurrences/progressions have occurred. The final analysis will be conducted when all 284 expected events have occurred.
  Defined as time from randomization to death due to melanoma. Death due to causes other than melanoma are not considered events for this analysis.
Time to development of new metastatic sites. | 3 interim analyses will be conducted when 75, 148, and 217 primary events have occurred. The final analysis will be conducted when all 284 expected events have occurred.
  This endpoint is defined as the time from randomization to disease recurrence at new metastatic sites in patients rendered disease-free by surgery, or time from randomization to the development of new metastatic sites of disease in patients in the best medical therapy group. Progression of existing lesions in the best medical therapy arm will not be considered an event for this endpoint.

CONTACTS AND LOCATIONS:
Overall Officials: Donald L. Morton, MD, Study Chair — Saint John's Cancer Institute
Locations (19):
- United States (15):
  - UC Davis Medical Center, Sacramento, California
  - John Wayne Cancer Institute, Santa Monica, California
  - Rush University, Chicago, Illinois
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Buffalo General Hospital, Buffalo, New York
  - Wake Forest University, Winston-Salem, North Carolina
  - Ohio State University Medical Center, Columbus, Ohio
  - Penn State Hershey Cancer Center, Hershey, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Geisinger Clinic, Wilkes-Barre, Pennsylvania
  - Main Line Health System, Wynnewood, Pennsylvania
  - Dallas Surgical Group, Dallas, Texas
  - UT Southwestern Medical Center at Dallas, Dallas, Texas
  - IHC Cancer Services Intermountain Healthcare, Murray, Utah
  - Huntsman Cancer Institute, Salt Lake City, Utah
- Princess Alexandra Hospital, Brisbane, Queensland, Australia
- Tel-Aviv Sourasky Medical Center, Tel Aviv, Israel
- Istituto Nazionale dei Tumori Napoli, Naples, Italy
- Univesitair Medisch Centrum Groningen, Groningen, Netherlands